CLINICAL TRIAL: NCT06568939
Title: A Phase 2, Open-Label, Randomized, Global Study of Three Telisotuzumab Vedotin Regimens in Subjects With Previously Treated c-Met Overexpressing, EGFR Wildtype, Locally Advanced/Metastatic Non-Squamous Non-Small Cell Lung Cancer
Brief Title: A Study to Assess Adverse Events and How Intravenously (IV) Infused Telisotuzumab Vedotin (ABBV-399) Moves Through the Body as a Monotherapy in Adult Participants With Previously Treated Non-Squamous Non-Small Cell Lung Cancer (NSCLC)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M25-274
Record Dates: First submitted 2024-08-22; First posted 2024-08-23 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; NSCLC; Telisotuzumab Vedotin; ABBV-399; TeliMET NSCLC-04
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — telisotuzumab vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Telisotuzumab Vedotin Dose A (Experimental): Participants will receive telisotuzumab vedotin dose A, as part of the 3 year study duration.
  Interventions: Drug: Telisotuzumab Vedotin
- Telisotuzumab Vedotin Dose B (Experimental): Participants will receive telisotuzumab vedotin dose B, as part of the 3 year study duration.
  Interventions: Drug: Telisotuzumab Vedotin
- Telisotuzumab Vedotin Dose C (Experimental): Participants will receive telisotuzumab vedotin dose C, as part of the 3 year study duration.
  Interventions: Drug: Telisotuzumab Vedotin

INTERVENTIONS:
Drug: Telisotuzumab Vedotin — Intravenous (IV) Infusion
  Other Names: ABBV-399

SUMMARY:
Cancer is a condition where cells in a specific part of body grow and reproduce uncontrollably. Non-small cell lung cancer (NSCLC) is a solid tumor, a disease in which cancer cells form in the tissues of the lung. The purpose of this study is to assess how safe telisotuzumab vedotin is in adult participants with NSCLC. Change in disease activity and adverse events will be assessed.

Telisotuzumab vedotin is an investigational drug being developed for the treatment of NSCLC. Participants will be randomly assigned a treatment of telisotuzumab vedotin in 1 of 3 arms at an 1:1:1 ratio. Each group receives intravenous (IV) infusion of telisotuzumab vedotin at different doses. Approximately 150 adult participants with c-Met overexpressing NSCLC will be enrolled in the study at approximately 70 to 80 sites worldwide.

Participants will receive IV telisotuzumab vedotin at 1 of 3 dose regimens as part of a 3 year study duration.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Projected life expectancy of at least 12 weeks.
* Must have c-Met overexpressing non-small cell lung cancer (NSCLC) as assessed by an AbbVie designated immunohistochemistry (IHC) laboratory
* Must have histologically or cytologically documented NSCLC that is locally advanced or metastatic.
* Must have a known epidermal growth factor receptor (EGFR) activating mutation status.
* Actionable alterations in genes other than EGFR are permitted.
* Must have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
* Must have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1.
* Must have received no more than 1 line of prior systemic cytotoxic chemotherapy in the locally advanced or metastatic setting, as stated in the protocol.
* Must have progressed on at least 1 line of prior therapy for locally advanced/metastatic NSCLC, as stated in the protocol.

Exclusion Criteria:

* Adenosquamous or neuroendocrine histology, or sarcomatoid features.
* Actionable EGFR activating mutations.
* Received prior c-Met-targeted antibodies, prior telisotuzumab vedotin, or prior antibody-drug conjugates either targeting c-Met or consisting of monomethylauristatin E.
* Received prior docetaxel therapy.
* Metastases to the central nervous system (CNS). Participants with CNS metastases are eligible only after adequate treatment (such as surgery or, radiotherapy, or drug therapy) is provided, as stated on the protocol.
* History of other malignancies except those stated in the protocol.
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan, as noted in the protocol.
* Unresolved clinically significant adverse event (AE) >= Grade 2 from prior anticancer therapy, except for alopecia or anemia. Participants with hormone deficiencies caused by prior anticancer therapy who are asymptomatic and on a stable dose of replacement hormone are eligible for study.
* Major surgery within 21 days prior to randomization.
* Clinically significant condition(s) including but not limited to those listed in the protocol.
* Clinically significant liver disease, including hepatitis, current alcohol abuse, or cirrhosis.
* Grade >= 2 edema or lymphedema.
* Grade >= 2 ascites or pleural effusion.
* Grade >= 2 neuropathy.
* Active uncontrolled bacterial or viral infection.
* Active corneal disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Treatment-Emergent Adverse Events (AE)s (Any-grade and Grade >= 2) | Up to Approximately 3 Years
  An AE is defined as any untoward medical occurrence, inappropriate participant management decision, unintended disease or injury or any untoward clinical signs (including an abnormal laboratory finding) in participants, users or other persons whether or not related to the investigational medical device.
Percentage of Participants with Treatment-Emergent Interstitial Lung Disease (ILD) | Up to Approximately 3 Years
  ILD is defined by ILD standardized MedDRA query (SMQ) (broad) per investigator and determined per adjudication (any-grade and Grade >= 2).
Percentage of Participants with Treatment-Emergent Peripheral Neuropathy | Up to Approximately 3 Years
  Peripheral neuropathy is defined by peripheral neuropathy SMQ (narrow) (any-grade and Grade >= 2)
Percentage of Participants with Treatment-Emergent Ocular Surface Disorders | Up to Approximately 3 Years
  Treatment-emergent ocular surface disorders defined by corneal epitheliopathy company MedDRA query (CMQ) (any-grade and Grade >= 2).
Percentage of Participants with Treatment-Emergent AEs Leading to Study Drug Discontinuation | Up to Approximately 3 Years
  An AE is defined as any untoward medical occurrence, inappropriate participant management decision, unintended disease or injury or any untoward clinical signs (including an abnormal laboratory finding) in participants, users or other persons whether or not related to the investigational medical device.
Percentage of Participants with Grade 5 Treatment-Emergent AEs | Up to Approximately 3 Years
  An AE is defined as any untoward medical occurrence, inappropriate participant management decision, unintended disease or injury or any untoward clinical signs (including an abnormal laboratory finding) in participants, users or other persons whether or not related to the investigational medical device.
Objective Response (OR) by Blinded Independent Central Review (BICR) | Up to Approximately 3 Years
  OR will be defined as achieving confirmed complete response (CR) or confirmed partial response (PR) based on response evaluation criteria in solid tumors (RECIST), version 1.1.

SECONDARY OUTCOMES:
Concentrations of Telisotuzumab Vedotin Conjugate in Serum | Up to 26 Weeks
  Concentrations of telisotuzumab vedotin conjugate in serum.
Concentrations of Monomethylauristatin E (MMAE) Payload in Plasma | Up to 26 Weeks
  Concentrations of MMAE payload in plasma.
Percentage of Participants with Antidrug Antibodies (ADAs) of Telisotuzumab Vedotin | Up to 26 Weeks
  Percentage of participants with ADAs of telisotuzumab vedotin.
Percentage of Participants with Neutralizing Antidrug Antibodies (nADAs) of Telisotuzumab Vedotin | Up to 26 Weeks
  Percentage of participants with nADAs of telisotuzumab vedotin.
Change in Selected items of the Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Cycle 1: Day 1, Day 8, Cycle 2 D1 and D1 of Every Even Cycle Thereafter, Through 3 Years
  The PRO-CTCAE is a patient-reported outcome measurement system developed to assess symptomatic toxicity in patients participating in cancer clinical trials. PRO-CTCAE includes 124 items representing 78 symptomatic toxicities drawn from the Common Terminology Criteria for Adverse Events (CTCAE). PRO-CTCAE items evaluate the symptom attributes of frequency, severity, interference, amount, presence/absence. All questions employ a 7-day recall period and are scored from 0 to 4 (or 0/1 for absent/present).
Change in GP5 item of the Functional Assessment of Cancer Therapy-General (FACT-G) | Cycle 1: Day 1, Day 8, Cycle 2 D1 and D1 of Every Even Cycle Thereafter, Through 3 Years
  The GP5 item ("I am bothered by side effects of treatment") of FACT-G is used to assess overall treatment tolerability in patients by assessing the overall side effect impact on participants.
Duration of Response (DoR) by BICR | Up to Approximately 3 Years
  DoR is defined for confirmed responders as the time from the participants' initial response (CR or PR) to the first occurrence of radiographic progression per RECIST v1.1 or death from any cause.
Progression-Free Survival (PFS) by BICR | Up to Approximately 3 Years
  PFS will be defined as the time from randomization to the first occurrence of radiographic progression based on RECIST version 1.1 or death from any cause.
Overall Survival (OS) | Up to Approximately 3 Years
  OS will be defined as the time from randomization to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (62):
- United States (34):
  - Ironwood Cancer & Research Center /ID# 276370, Chandler, Arizona
  - University of Arkansas for Medical Sciences /ID# 272923, Little Rock, Arkansas
  - Valkyrie Clinical Trials /ID# 271322, Los Angeles, California
  - Yale New Haven Hospital /ID# 271584, New Haven, Connecticut
  - Cancer Specialists of North Florida - Jacksonville - AC Skinner Parkway /ID# 270899, Jacksonville, Florida
  - Ocala Oncology Center /ID# 273697, Ocala, Florida
  - Comprehensive Hematology Oncology /ID# 270422, St. Petersburg, Florida
  - Florida Cancer Specialists - North /ID# 271995, St. Petersburg, Florida
  - Florida Cancer Specialists - East /ID# 271993, West Palm Beach, Florida
  - University Cancer & Blood Center /ID# 270969, Athens, Georgia
  - Northwest Georgia Oncology Centers /ID# 275374, Marietta, Georgia
  - Memorial University Medical Center /ID# 272467, Savannah, Georgia
  - Kaiser Permanente Moanalua Medical Center /ID# 272916, Honolulu, Hawaii
  - University of Illinois Hospital and Health Sciences System /ID# 275345, Chicago, Illinois
  - Illinois Cancer Specialists /ID# 274678, Niles, Illinois
  - Springfield Clinic - First /ID# 272576, Springfield, Illinois
  - NHO - Nebraska Hematology-Oncology /ID# 272970, Lincoln, Nebraska
  - Nebraska Cancer Specialists - Omaha - Wright Street /ID# 271527, Omaha, Nebraska
  - Renown Regional Medical Center /ID# 273535, Reno, Nevada
  - Astera Cancer Care /ID# 272359, East Brunswick, New Jersey
  - Montefiore Medical Center /ID# 277169, The Bronx, New York
  - Clinical Research Alliance - Westbury /ID# 270455, Westbury, New York
  - FirstHealth of the Carolinas- Speciality Center /ID# 272924, Pinehurst, North Carolina
  - Mercy Health - Perrysburg Cancer Center /ID# 270536, Perrysburg, Ohio
  - Genesis Healthcare System /ID# 273361, Zanesville, Ohio
  - Guthrie Robert Packer Hospital /ID# 270316, Sayre, Pennsylvania
  - Cancer Care Associates Of York /ID# 270971, York, Pennsylvania
  - Saint Francis Cancer Center - Greenville /ID# 276368, Greenville, South Carolina
  - SCRI Oncology Partners /ID# 270162, Nashville, Tennessee
  - Texas Oncology - Northeast Texas /ID# 272000, Tyler, Texas
  - Community Cancer Trials Of Utah /ID# 276598, Ogden, Utah
  - Virginia Cancer Specialists - Fairfax /ID# 272004, Fairfax, Virginia
  - Medical Oncology Associates - Spokane /ID# 277172, Spokane, Washington
  - Northwest Medical Specialties Tacoma /ID# 270534, Tacoma, Washington
- China (8):
  - Beijing Chest Hospital, Capital Medical University /ID# 271935, Beijing, Beijing Municipality
  - Affiliated Cancer Hospital of Guangxi Medical University /ID# 271931, Nanning, Guangxi
  - Henan Cancer Hospital /ID# 271927, Zhengzhou, Henan
  - Union Hospital - Tongji Medical College /ID# 271668, Wuhan, Hubei
  - The First Affiliated Hospital of Nanchang University /ID# 271666, Nanchang, Jiangxi
  - The First Affiliated Hospital of Xi'an Jiaotong University /ID# 271928, Xi'an, Shaanxi
  - Linyi Cancer Hospital /ID# 272068, Linyi, Shandong
  - Cancer Hospital Affliated to Xinjiang Medical University /ID# 271933, Ürümqi, Xinjiang
- Israel (4):
  - Meir Medical Center /ID# 270071, Kfar Saba, Central District
  - Rambam Health Care Campus- Haifa /ID# 270078, Haifa
  - Shaare Zedek Medical Center /ID# 270095, Jerusalem
  - Rabin Medical Center. /ID# 270087, Petah Tikva
- Japan (8):
  - Nagoya University Hospital /ID# 277010, Nagoya, Aichi-ken
  - Hokkaido University Hospital /ID# 277014, Sapporo, Hokkaido
  - Kobe Minimally Invasive Cancer Center /ID# 277469, Kobe, Hyōgo
  - Kitasato University Hospital /ID# 277012, Sagamihara-shi, Kanagawa
  - Sendai Kousei Hospital /ID# 277023, Sendai, Miyagi
  - University of Miyazaki Hospital /ID# 277020, Miyazaki, Miyazaki
  - Fujieda Municipal General Hospital /ID# 277025, Fujieda, Shizuoka
  - Wakayama Medical University Hospital /ID# 276997, Wakayama, Wakayama
- Serbia (6):
  - Institute for Oncology and Radiology of Serbia /ID# 270561, Belgrade, Beograd
  - University Clinical Center Serbia /ID# 270808, Belgrade, Beograd
  - Clinical Hospital Center - Bežanijska Kosa /ID# 270558, Belgrade, Beograd
  - University Clinical Center Nis /ID# 270557, Niš, Nisavski Okrug
  - Institute For Pulmonary Diseases Of Vojvodina /ID# 270559, Kamenitz, Sremski Okrug
  - University Clinical Center Kragujevac /ID# 275773, Kragujevac, Sumadijski Okrug
- Singapore (2):
  - National Cancer Centre Singapore /ID# 271499, Singapore, Central Singapore
  - National University Hospital /ID# 271700, Singapore

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M25-274